CLINICAL TRIAL: NCT04205149
Title: Post-Operative Recovery After Cesarean Hysterectomy Using the Enhanced Recovery After Surgery (ERAS) Pathway
Brief Title: Enhanced Recovery After Cesarean Hysterectomy
Status: Withdrawn | Type: Observational
Why Stopped: research staff leading project left institute
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Ai-ris Collier, Principal Investigator, Beth Israel Deaconess Medical Center
Other Study IDs: 2019P000821
Record Dates: First submitted 2019-09-30; First posted 2019-12-19 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Post-operative Recovery for Cesarean Hysterectomy Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-ERAS implementation arm
- Post-ERAS implementation arm
  Interventions: Other: ERAS post-operative pathway

INTERVENTIONS:
Other: ERAS post-operative pathway — ERAS Pathway
  Groups: Post-ERAS implementation arm

SUMMARY:
The enhanced recovery after surgery (ERAS) pathway is a well-described evidence-based protocol to optimize patient post-operative recovery. Patients undergoing cesarean hysterectomies are a unique surgical population. These procedures are most commonly performed for patients with placenta accreta spectrum or severe postpartum hemorrhage. In recent studies examining the effectiveness of the ERAS pathway, post-operative cesarean patients experienced decreased average inpatient opioid exposure without an increase in pain scores, early mobilization and nutrition targets without increases in adverse outcomes after program implementation. Post-operative hysterectomy patients with gynecologic indications experienced shorter lengths of stay and decreased opioid consumption. Additionally, patients have significantly higher satisfaction scores. The investigators suspect that this population may also benefit similarly.

This research is a pre- and post- study to assess and describe surgical outcomes and parameters surrounding patients' post-operative recovery and experience before and after the ERAS pathway is implemented at a high volume placenta accreta spectrum Center of Excellence.

DETAILED DESCRIPTION:
The enhanced recovery after surgery (ERAS) pathway has emerged as an evidence-based protocol to optimize patient post-operative recovery. It utilizes multimodal analgesia to decrease narcotic use and promote streamlined patient-centered care that helps to reduce blood loss, expedite patients' return to baseline function, and prepare patient expectations around surgery. This pathway has been well studied in several surgical populations, including gynecologic (post hysterectomy) and obstetric (post cesarean) patients.

Patients undergoing cesarean hysterectomies are a unique surgical population. These procedures are most commonly performed for patients with placenta accreta spectrum or severe postpartum hemorrhage. Ideally, women with suspected placenta accreta spectrum diagnosed antenatally should be delivered at a level III or IV center with placenta accreta spectrum Centers of Excellence accreditation to improve outcomes. With the rates of placenta accreta spectrum increasing, these Centers of Excellence could consider applying principles of the ERAS pathway to the operative management of these patients. Other populations have seen decreases in opioid use, quicker baseline recovery, shorter hospital stays and overall improved patient satisfaction with the use of the ERAS pathway.

In recent studies examining the effectiveness of the ERAS pathway, post-operative cesarean patients experienced decreased average inpatient opioid exposure without an increase in pain scores, early mobilization and nutrition targets without increases in adverse outcomes after program implementation. Post-operative hysterectomy patients with gynecologic indications experienced shorter lengths of stay and decreased opioid consumption. Additionally, patients have significantly higher satisfaction scores. The investigators suspect that this population may also benefit similarly.

This research is a pre- and post- study to assess and describe surgical outcomes and parameters surrounding patients' post-operative recovery and experience before and after the ERAS pathway is implemented at a high volume placenta accreta spectrum Center of Excellence.

The study design involves a retrospective analysis of variables related to postpartum recovery. The primary outcome will be oral morphine equivalents as a proxy for narcotic use in the first 72 hours post-operatively, comparing pre- to post-ERAS implementation. Investigators will also collect data on pain scores, time to ambulation, time to foley catheter removal and first void, and length of stay. Investigators will also collect data on post-operative complications including surgical site infection, urinary tract infection, transfusion, unplanned return to OR, pneumonia, pulmonary embolism, unplanned intubation, cardiac arrest, readmission within 30 days, sepsis, and death within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Underwent a cesarean hysterectomy at Beth Israel Deaconess Medical Center

Exclusion Criteria:

* Patient records not accessible at Beth Israel Deaconess Medical Center

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing cesarean hysterectomy at Beth Israel Deaconess Medical Center
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Oral morphine equivalents | Until study completion, expected 2 years
  Oral morphine equivalent use during first 72 hours after surgery

SECONDARY OUTCOMES:
Pain scores | Until study completion, expected 2 years
  Likert scale 0-10 (0=no pain, 10=most pain) during first 72 hours after surgery
Time to ambulation | Until study completion, expected 2 years
  Hours from surgery to first ambulation
Time to urinary foley removal | Until study completion, expected 2 years
  Hours from surgery to foley catheter removal
Length of stay | Until study completion, expected 2 years
  Days of inpatient hospitalization after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No